CLINICAL TRIAL: NCT06126926
Title: Mobilizing Evidence Into Tertiary Prevention of Child Sexual Abuse: A Pilot Study
Brief Title: Tertiary Prevention of Child Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FMCH-2023-32331
Record Dates: First submitted 2023-10-16; First posted 2023-11-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Child Sexual Abuse
MeSH Terms: interventions — Psychotherapy, Group; Therapeutics

STUDY DESIGN:
Intervention Model Description: Random assignment clinical trial. Participants are randomly assigned to the intervention group or treatment as usual.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 32-week group therapy
  Interventions: Behavioral: group therapy
- Control group (Active Comparator): Treatment as Usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: group therapy — 32 weeks of group therapy
  Arms: Intervention arm
Other: Treatment as usual — Control participants remain in their current placement and may be eligible for a number of services offered to inmates to facilitate rehabilitation and planning for release to the community, including sexual offender treatment. MnDOC's sexual offender treatment is a two to three year program, thus most of our control subjects will not have enough time remaining on their sentences to complete such treatment. However, a number of them may participate in MnDOC's current program.
  Arms: Control group

SUMMARY:
This is a feasibility study designed to inform the development of a multinational study of the effectiveness of a tertiary prevention program for child sexual abuse. This study targets adult men who have engaged in child sexual abuse, and will be implemented within the Minnesota Department of Corrections. Data will include measures of the implementation process, short-terms changes in criminogenic factors, and staff and participant factors that could influence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 or older
* Serving time in MnDOC facilities for Criminal Sexual Conduct in the first, second, or third degree, whose victims were less than 14 years old
* Individuals assigned moderate to high risk to reoffend as determined upon entrance to the Minnesota Correctional System by the DOC Risk Assessment/Community Notification Unit."

Exclusion Criteria:

* Diagnosed with an active, uncontrolled major mental disorder (e.g. bi-polar, schizophrenia, schizoaffective disorder, major depression with psychotic features)
* Unable to read English at the 5th grade level
* Unable to speak English
* IQ of less than 85 as measured by standard intelligence tests
* Diagnosis of intellectual disability
* Engaged in violent behavior while incarcerated, as indicated by disciplinary actions and/or segregation within 60 days of intake"

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes, the current study includes only men, as the intervention is designed for men who have perpetrated child sexual abuse.
Enrollment: 10 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Violence Risk Scale-Sexual Offense Version (VRS:SO) | 7 days post-intervention
  Clinician rating scale. 24-items measuring likelihood of sexual offense recidivism using a 4 point scale.
Coping Using Sex Inventory (CUSI) | 7 days post-intervention
  Self-report scale. 16 items measuring consensual, non-consensual, and child-focused sexual coping strategies using a 5-point scale
Compulsive Sexual Behavior Inventory-13 (CSBI-13) | 7-days post-intervention
  Self-report scale. 13 item scale measuring the presence of compulsive sexual behaviors on a 5- point scale.
Types of Jealousy Scale (3 subscales; reactive, preventive, and anxious jealousy) | 7 days post-intervention
  Self-report scale. 15 items measuring the intensity of reactive jealousy, experience and use of preventive jealousy, and frequency of anxious jealousy on a 5-point scale.
Faith in People Scale | 7 days post-intervention
  Self-report scale. 5 item scale measuring attitudes toward human nature. Two forced- choice items and three agreement/disagreement items.
Trust in People Scale (Survey Research Center) | 7 days post-intervention
  Self-report scale. 3 item scale measuring perception of general trustworthiness of others.
Aggression Questionnaire (AQ; Buss &amp) - Physical Aggression, Verbal Aggression, and Anger Subscales ONLY | 7 days post-intervention
  Self-report scale. 21 items throughout the 3 subscales measuring how characteristic physical aggression, verbal aggression, and anger-related behaviors are for respondents on a 7 point scale.
Revised UCLA Loneliness Scale (R-UCLA) | 7 days post-intervention
  Self-report scale. 20 items measuring subjective feelings of loneliness and social isolation on a 4 point scale.
Self-Critical Rumination Scale (SCRS) | 7 days post-intervention
  Self-report scale. 10 items measuring self- criticism on a 4 point scale.
External/Internal Shame Scale - Sense of Isolation/Exclusion Subscale ONLY (EISS) | 7 days post-intervention
  Self-report scale. Measures perceived sense of exclusion and being isolated or misunderstood by people on a 5 point scale.
Children and Sex Questionnaire Emotional Congruence Scale (CSQ:ECWC) | 7 days post-intervention
  Self-report scale. 15 item scale measuring emotional congruence with children on a 5 point scale.
The Openness to Men and Women Scales (OPM, OPWO) | 7 days post-intervention
  Self-report scale. 18 items assessing openness to intimacy with women and men on a 4 point scale.
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | 7 days post-intervention
  Self-report scale. 18 items measuring problems with emotion regulation including subscales for strategies, non-acceptance, impulse, goals, awareness, and clarity on a 5 point scale.
Coping Strategy Indicator (CSI) | 7 days post-intervention
  Self-report scale. 33 items measuring adaptive and maladaptive coping strategies (avoidance, problem-solving, social support seeking) on a 3 point scale.
Aggression Inventory (AI)- Impulsive, Impatient, and Avoid subscales ONLY | 7 days post-intervention
  Self-report scale. 22 item scale measuring perceptions and use of aggressive behaviors for men a women on a 5 point scale.

SECONDARY OUTCOMES:
Group Climate Questionnaire - Short Form (GCQ-5) | Every 14 days for first two months, than every four weeks for next four months
  Self-report scale. 12 items measuring group perceptions of the group therapeutic environment on a 7 point scale.
Curative Climate Instrument (CCI) | Every 14 days for first two months, than every four weeks for next four months
  Self-report scale. 14 items measuring specific change processes perceived as helpful to individual group members (catharsis, insight, and cohesiveness) on a 5 point scale.
Treatment Motivation Questionnaire-Revised (TMQ-R) | Every 14 days for first two months, than every four weeks for next four months
  Self-report scale. 23 items measuring internal and external reasons for participating in treatment, motivations relating to connecting and sharing with others, and clients' potential lack of confidence in treatment on a 7 point scale.
Therapeutic Agency Inventory (TAI) | Every 14 days for first two months, than every four weeks for next four months
  Self-report scale. 15 items measuring clients' experience of agency in making positive change and ability to take an active role in their therapy on a 5 point scale.
Relationship Questionnaire (RQ) | Every 14 days for first two months, than every four weeks for next four months
  Self-report scale. 4 items measuring adult attachment style on a 7 point scale.
Working Alliance Inventory - Short Form (WAI- SR) | Every 14 days for first two months, than every four weeks for next four months
  Self-report scale. 12 items measuring three domains of the therapeutic alliance: goals, tasks, and bond on a 5 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miner, Ph.D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States